CLINICAL TRIAL: NCT07222657
Title: Phase 2 Randomized Trial Of Liquid Nitrogen Spray Cryotherapy Prior To Neoadjuvant Systemic Therapy In Locally Advanced Esophageal Adenocarcinoma
Brief Title: Liquid Nitrogen Spray Cryotherapy Prior to Neoadjuvant Systemic Therapy in Esophageal Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Salgi Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE14225
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Adenocarcinoma; Esophageal Cancer
Keywords: Liquid Nitrogen Spray Cryotherapy; LNSC
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid Nitrogen Spray Cryotherapy (LNSC) + Standard of care chemotherapy (Experimental): Participants will receive a standard of care chemotherapy, neoadjuvant FLOT +/- durvalumab WITH LNSC.
  Interventions: Other: Standard of care chemotherapy; Procedure: LNSC
- Standard of care chemotherapy (Other): Participants will receive a standard of care chemotherapy, neoadjuvant FLOT +/- durvalumab WITHOUT LNSC.
  Interventions: Other: Standard of care chemotherapy

INTERVENTIONS:
Other: Standard of care chemotherapy — Participants will receive neoadjuvant therapy per FLOT protocol +/- Durvalumab for up to 6 cycles. Each cycle is two weeks.
  The FLOT protocol is a standard of care protocol involving chemotherapy before and after esophagectomy with fluorouracil, leucovorin, oxaliplatin, and docetaxel.
  Durvalumab is administered intravenously (IV) and dosed at 1500 milligrams (mg). It is given on Day 1 of each cycle.
Procedure: LNSC — LNSC will be administered via endoscopy. LNSC will be performed with liquid nitrogen (<5 psi) at 25 watts using a cryotherapy catheter passed through the working channel of the endoscope. Up to three cycles of 20 to 40 seconds of cryotherapy will be administered and each directed at the bulkiest aspect of the tumor. During each cycle, a surface area of approximately 2 to 3 cm2 is targeted, and up to three sites are targeted during each session.
  Participants will receive two sessions of LNSC. The first will be upon entry into the study. The second will be 1-2 weeks after the first session.
  Arms: Liquid Nitrogen Spray Cryotherapy (LNSC) + Standard of care chemotherapy

SUMMARY:
This research study is for people who have locally advanced esophageal adenocarcinoma and are expected to receive chemotherapy. The purpose of this study is to compare the effectiveness of Liquid Nitrogen Spray Cryotherapy (LNSC) in addition to chemotherapy versus chemotherapy alone in the treatment of esophageal adenocarcinoma. LNSC is an FDA approved device that works by using liquid nitrogen to rapidly cool cancerous tissue causing cell damage. Participants in this study will be randomly assigned to either the "LNSC group" or the "No-LNSC group." Participants in the "LNSC group" will undergo 2 sessions of LNSC through an upper endoscopy. Participants in the "No-LNSC group," may undergo an endoscopy if needed for symptoms such as difficulty swallowing. Participation in the research will last about 4 months.

DETAILED DESCRIPTION:
People with locally advanced esophageal adenocarcinoma (a type of cancer in the esophagus) often have trouble swallowing because of the tumor's size and spreading to nearby areas. Doctors diagnose and stage the cancer using upper endoscopy, cross-sectional imaging, and endoscopic ultrasonography. Management of locally advanced esophageal adenocarcinoma usually involves more than one type of therapy. Treatment often includes chemotherapy and surgical resection in operable cases. Studies show that complete response (CR) rates are low with neoadjuvant therapy for esophageal cancer. For example, pathologic CR (PCR) to neoadjuvant chemoradiation (CROSS) occurs in only 25-30% of people with locally advanced esophageal cancer. CR strongly correlates with overall survival in esophageal cancer. Therefore, additional neoadjuvant therapies/regimens are required to improve survival for people with this type of cancer.

Liquid nitrogen spray cryotherapy (LNSC) is a treatment for destroying abnormal tissue in Barrett's esophagus (BE) and esophageal cancer (EC). During LNSC, liquid nitrogen is sprayed through a thin tube that is passed through the working channel of a gastroscope. Liquid nitrogen rapidly cools neoplastic tissue to extremely low temperatures (-78°C to -196°C), causing intracellular ice formation. The freezing process leads to cell membrane rupture, protein denaturation, and microvascular thrombosis. This leads to cell death (necrosis) of the abnormal tissue.

Liquid Nitrogen Spray Cryotherapy (LNSC) may increase CR by boosting the body's immune response, which helps to fight and destroy the tumor cells. It is FDA-approved for debulking esophageal cancer. In a prospective multi-center study, it was found that LNSC caused minimal side effects and improves Quality of Life (QoL) in people with esophageal cancer that cannot have surgery and who were receiving systemic therapy. In a pilot clinical trial, it was found that LNSC resulted in a long-term CR rate of 56% when a single session of LNSC was administered prior to CROSS. When compared to matched participants who received CROSS alone, immune cells that fight tumor cells multiplied more frequently with LNSC + CROSS. Investigators then conducted a neoadjuvant LNSC dose frequency escalation trial. There was improved QoL and no severe (grade 3) side effects with two sessions of neoadjuvant LNSC. Consistent with our prior study, 64% of people who completed at least two sessions of LNSC had a clinical complete CR (CCR) after CROSS. These findings support the need for a larger study to investigate whether adding LNSC can improve treatment of locally advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults with locally advanced EAC who are expected to receive FLOT +/-Durvalumab will be eligible to participate.
* Locally advanced esophageal cancer is defined as TNM stages T1N+M0 or T2-T4aNanyM0, as defined by endoscopic ultrasound (EUS) and PET-CT.

Exclusion Criteria:

* Inability to pass the orogastric decompression tube into the stomach
* Coagulopathy (INR > 2 or platelet count < 50,000 per cubic millimeter)
* Inability to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Risk of thrombosis is determined to be too high to hold anti-platelets (other than aspirin) or anticoagulants prior to the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rates | At treatment discontinuation, up to 12 weeks
  CR is defined as the absence of tumor on re-staging scans and explant or mucosal biopsies (if applicable).

SECONDARY OUTCOMES:
Change in minimal residual disease (MRD) | Week 4 of chemotherapy, 2-4 weeks post-chemotherapy (up to 16 weeks)
  MRD is defined using the Signatera assay as any detectable circulating tumor DNA (ctDNA)
Overall survival (OS) | 1 year
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death from any cause.
Change in systemic immune response | Baseline, 4 weeks post-chemotherapy, up to 16 weeks
  Systemic immune response will be measured through cellular immune profiling (e.g., CD4+, CD8+, cytotoxic T cells, FOXP3+ regulatory T cells) via centralized flow cytometry.
Change in dysphagia | Baseline, up to 2 weeks
  Dysphagia is measured by a Dysphagia Questionnaire containing 5 questions. Participants answer 3 questions with yes/no answer choices that refer to if they have had trouble swallowing. Participants answer 1 question regarding severity of dysphagia with 4 answer choices ranging from "Doesn't bother me at all" to "Very severe." Participants answer 1 question regarding frequency of dysphagia with answer choices ranging from "None" to "Unable to eat." Participants answer 1 question regarding the type of items that have trouble swallowing with answer choices being "Both solids and liquids," "Solid foods only," or "Liquids only." Answers are qualitatively assessed for severity and frequency of dysphagia.
Change in quality of life (QoL) | Baseline, up to 2 weeks
  QoL is measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Oesophageal Cancer 18 (EORTC QLC - OES18). This is an 18-item questionnaire, where participants rate their quality of life on a 4-point Likert scale ranging from 1 (Not at All) to 4 (Very much). Greater scores indicate lower quality of life.
LNSC-related adverse events | 30 days post-treatment, up to 20 weeks
  Incidence of LNSC-related adverse events will be measured by CTCAE version 5.0 or 6.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tilak Shah, MD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 6 months of study completion
Access Criteria: Public

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Kachaamy T, Sharma N, Shah T, Mohapatra S, Pollard K, Zelt C, Jewett E, Garcia R, Munsey R, Gupta S, Rojas-DeLeon M, Gupta D, Kaul V, Pannala R, Vashi P. A prospective multicenter study to evaluate the impact of cryotherapy on dysphagia and quality of life in patients with inoperable esophageal cancer. Endoscopy. 2023 Oct;55(10):889-897. doi: 10.1055/a-2105-2177. Epub 2023 Jun 2. PMID 37268010
- [Background] Shah T, Kushnir V, Mutha P, Majhail M, Patel B, Schutzer M, Mogahanaki D, Smallfield G, Patel M, Zfass A. Neoadjuvant cryotherapy improves dysphagia and may impact remission rates in advanced esophageal cancer. Endosc Int Open. 2019 Nov;7(11):E1522-E1527. doi: 10.1055/a-0957-2798. Epub 2019 Oct 31. PMID 31681831
- [Background] Shah T, Koblinski J, Boothello R, Haneefa SM, Massey HD, Patel BB. Changes in Local Tumor Immune Microenvironment with Neoadjuvant Cryotherapy and Chemoradiation for Locally Advanced Esophageal Cancer. Foregut. 2024;0(0).
- [Background] Shah T, Spataro J, Mutha P et al. Phase 1 dose frequency escalation study of neoadjuvant cryotherapy in locally advanced esophageal cancer. Gastrointestinal Endoscopy, Volume 97, Issue 6, AB1106 - AB1107.